CLINICAL TRIAL: NCT06607523
Title: The Gut-Brain Axis During Neurorehabilitation; Prebiotic Treatment to Alter the Gut Microbiome and Neurologic Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: Moody Neurorehabilitation Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-0237
Record Dates: First submitted 2024-09-03; First posted 2024-09-23 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Brain Injuries
Keywords: Brain Injury; Neurorehabilitation; Fatigue; Cognition
MeSH Terms: conditions — Brain Injuries; Fatigue | interventions — Inulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Community Controls (No Intervention): Community Control subjects will not receive intervention.
- Brain Injury Patients - no intervention (No Intervention): Brain injury patients receiving residential standard of care post-acute neurorehabilitation.
- Brain Injury Patients - inulin intervention (Active Comparator): Brain injury patients receiving residential standard of care post-acute neurorehabilitation plus 42 days of daily oral inulin supplementation (4g 2x daily).
  Interventions: Dietary Supplement: Inulin

INTERVENTIONS:
Dietary Supplement: Inulin — Inulin, 4g twice daily for 42 days
  Arms: Brain Injury Patients - inulin intervention

SUMMARY:
The aim of this study is to characterize the microbiome of patients undergoing post-acute residential neurorehabilitation compared to community controls and to determine if a dietary fiber, Inulin, can create a shift in the microbiome leading to changes in fatigue and cognition.

DETAILED DESCRIPTION:
The investigative research team previously described Brain Injury Associated Fatigue and Altered Cognition (BIAFAC) as a treatable syndrome that occurs in a subset of patients following traumatic brain injury (TBI). In addition to fatigue and brain fog, BIAFAC patients have altered growth hormone (GH) secretion, reduced serum amino acid levels, and an altered (dysbiotic) gut microbiome. GH treatment dramatically improves patient symptoms but is not curative; symptoms return when GH treatment ends and the associated gut dysbiosis is not corrected. In preliminary work with mouse models created using human fecal transplants from clinical BIAFAC subjects, transplanting the dysbiotic gut bacteria from BIAFAC patients alone caused fatigue, altered cognition, and dysregulated GH secretion without any trauma or head injury. These mouse models indicate that gut dysbiosis has a causative role in the development of BIAFAC by triggering both altered GH secretion and neurologic symptoms. In this clinical trial a dietary fiber, Inulin, will be administered to patients undergoing neurorehabilitation after brain injury to create a shift in their microbiome.

Specific Aims

Aim 1. Identify differences in blood and fecal microbiome biomarkers of neurorehabilitation patients.

Specific Aim 1a. Identify differences in blood and fecal microbiome biomarkers between patients entering an inpatient post-acute neurorehabilitation program and community controls.

Specific Aim 1b. Identify correlations between biomarkers (blood and fecal microbiome), demographics (e.g. age, sex), and clinical factors (e.g. medical history) of post-acute neurorehabilitation patients.

Specific Aim 1c. Document longitudinal change in blood and fecal microbiome biomarkers of patients during inpatient post-acute neurorehabilitation.

Aim 2. Determine the effect of dietary inulin supplement on patients undergoing post-acute neurorehabilitation.

Specific Aim 2a. Determine how dietary inulin supplementation impacts the gut microbiome profile and function in brain injury patients during inpatient post-acute neurorehabilitation.

Specific Aim 2b. Determine if dietary inulin supplementation affects fatigue and cognition in patients during inpatient post-acute neurorehabilitation.

Aim 3. Determine if short-term early intervention dietary inulin supplementation during post-acute neurorehabilitation affects longer-term patient-reported outcomes.

ELIGIBILITY:
Brain Injury Patients

Inclusion

* Ages 18 and above
* Admitted to Moody Neurorehabilitation Institute for care
* Less than 6 months post-injury
* English speaking
* Must be able to eat and drink by mouth
* Willing and able to comply with study procedures
* Willing and able to provide consent (with LAR if needed)

Exclusion

* Significant heart, liver, kidney, blood or respiratory disease
* HIV, Hepatitis B or Hepatitis C
* Pregnancy or becoming pregnant during the study
* History of inflammatory bowel disease
* History of celiac disease
* Active diverticular disease
* Known allergy to study agent
* Any medical condition that, in the opinion of the investigator, would place the subject at increased risk for participation

Community Control Subjects

Inclusion

* Ages 18 and above
* Have a family member who is admitted to Moody Neurorehabilitation Institute for care OR is working at Moody Neurorehabilitation Institute
* English speaking
* Willing and able to comply with study procedures
* Willing and able to provide consent
* FACs score ≤ 50

Exclusion

* Trauma to head in last 6 months
* Stroke in last 6 months
* Significant heart, liver, kidney, blood or respiratory disease
* HIV, Hepatitis B or Hepatitis C
* Pregnancy or becoming pregnant during the study
* History of inflammatory bowel disease
* History of celiac disease
* Active diverticular disease
* Any medical condition that, in the opinion of the investigator, would place the subject at increased risk for participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Quantify absolute abundance of gut microbiome using metagenomic analysis at baseline | baseline
  Metagenomic analysis using a custom PCR array will be performed on stool samples to identify associated changes in microbiome absolute abundance at the genus and species level.
Quantify absolute abundance of gut microbiome using metagenomic analysis after 42 days of inulin supplementation | 42 days inulin treatment
  Metagenomic analysis using a custom PCR array will be performed on stool samples to identify associated changes in microbiome absolute abundance at the genus and species level.
Quantify absolute abundance of gut microbiome using metagenomic analysis at 3 months of discontinuation of inulin | 3 months of discontinuation of inulin
  Metagenomic analysis using a custom PCR array will be performed on stool samples to identify associated changes in microbiome absolute abundance at the genus and species level.
Quantify absolute abundance of gut microbiome using metagenomic analysis at 6 months of discontinuation of inulin | 6 months of discontinuation of inulin
  Metagenomic analysis using a custom PCR array will be performed on stool samples to identify associated changes in microbiome absolute abundance at the genus and species level.
Fold change in relative abundance of gut microbiome using metatranscriptomic analysis from baseline to 42 days of inulin treatment | From baseline to 42 days of inulin treatment
  Metatranscriptomic analysis using a RNA seq will be performed on stool samples to identify associated fold changes in which genes are turned on and off.
Fold change in relative abundance of gut microbiome using metatranscriptomic analysis from baseline to 3 months after discontinuation of inulin treatment | From baseline to 3 months after discontinuation of inulin treatment
  Metatranscriptomic analysis using a RNA seq will be performed on stool samples to identify associated fold changes in which genes are turned on and off.
Fold change in relative abundance of gut microbiome using metatranscriptomic analysis from baseline to 6 months after discontinuation of inulin treatment | From baseline to 6 months after discontinuation of inulin treatment
  Metatranscriptomic analysis using a RNA seq will be performed on stool samples to identify associated fold changes in which genes are turned on and off.

SECONDARY OUTCOMES:
Fatigue and Cognition as measured by the Fatigue and Altered Cognition Scale at baseline | baseline
  The Fatigue and Altered Cognition Scale (FACS) is a joint project from University of Texas Medical Branch and Texas A&M University. The FACS is a 20 question assessment designed to access perceived fatigue and cognition.
  There are 2 subscales used to calculate a total score. The subscales are: Fatigue and Altered Cognition. The total score is calculated by adding the subscales together. The range of the total score is 0-100, with a higher score indicating more fatigue and altered cognition.
Fatigue and Cognition as measured by the Fatigue and Altered Cognition Scale after 42 days of inulin treatment | 42 days of inulin treatment
  The Fatigue and Altered Cognition Scale (FACS) is a joint project from University of Texas Medical Branch and Texas A&M University. The FACS is a 20 question assessment designed to access perceived fatigue and cognition.
  There are 2 subscales used to calculate a total score. The subscales are: Fatigue and Altered Cognition. The total score is calculated by adding the subscales together. The range of the total score is 0-100, with a higher score indicating more fatigue and altered cognition.
Fatigue and Cognition as measured by the Fatigue and Altered Cognition Scale at 3 months after discontinuation of inulin | 3 months discontinuation of inulin
  The Fatigue and Altered Cognition Scale (FACS) is a joint project from University of Texas Medical Branch and Texas A&M University. The FACS is a 20 question assessment designed to access perceived fatigue and cognition.
  There are 2 subscales used to calculate a total score. The subscales are: Fatigue and Altered Cognition. The total score is calculated by adding the subscales together. The range of the total score is 0-100, with a higher score indicating more fatigue and altered cognition.
Fatigue and Cognition as measured by the Fatigue and Altered Cognition Scale at 6 months discontinuation of inulin | 6 months discontinuation of inulin
  The Fatigue and Altered Cognition Scale (FACS) is a joint project from University of Texas Medical Branch and Texas A&M University. The FACS is a 20 question assessment designed to access perceived fatigue and cognition.
  There are 2 subscales used to calculate a total score. The subscales are: Fatigue and Altered Cognition. The total score is calculated by adding the subscales together. The range of the total score is 0-100, with a higher score indicating more fatigue and altered cognition.

CONTACTS AND LOCATIONS:
Overall Officials: Randall Urban, MD, Principal Investigator — University of Texas; Ana Durand, MD, Study Director — Moody Neurorehabilitation Institute
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No